CLINICAL TRIAL: NCT03933774
Title: PHNA, Efficacy of Tretinoin Cream on Post-phototherapy Hyperpigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Min Bae, Department of Dermatology, St. Vincent's Hospital, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VC18MESI0278
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tretinoin 0.05% cream group (Experimental): Tretinoin 0.05% cream 25g for 1 month, applied on the half side of the face after randomization, once a day every night
  Interventions: Drug: Tretinoin 0.05% cream; Drug: Placebo cream
- Placebo (Placebo Comparator): PHYSIOGEL Daily Moisture Therapy Creme 150ml for 1 month, applied on the other half side of the face once a day every night
  Interventions: Drug: Tretinoin 0.05% cream; Drug: Placebo cream

INTERVENTIONS:
Drug: Tretinoin 0.05% cream — Stieva-A Cream 0.05%, 25g, GSK
Drug: Placebo cream — Physiogel Daily Mositure Therapy Facial cream, 150mL, Stiefel

SUMMARY:
A randomized controlled split-face pilot study was planned to investigate the preventive effect of tretinoin 0.05% cream on hyperpigmentation during phototherapy in patients with vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a chronic depigmentation disorder characterized by well-demarcated white macules and patches, reflecting selective melanocyte destruction. Hyperpigmentation at the treated areas is one of the limitations of phototherapy. Topical tretinoin (retinoic acid) has been well established to be effective for skin pigmentary disorders including melasma. This study aims to investigate the preventive effect of topical tretinoin on hyperpigmentation during phototherapy. A randomized controlled trial based on split-face was planned. The left/right face will be randomized to either tretinoin or placebo cream treatment groups. All lesions will be treated using phototherapy twice weekly for a total of 12-week period. The degree of repigmentation will be assessed as % from baseline by using a computer program every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 19
* A patient with stable non-segmental vitiligo
* A patient with symmetrical vitiligo lesions on face
* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it.
* A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* Age: lower than 20
* A pregnant or lactating patient
* A patient with active or spreading vitiligo
* A patient who cannot understand the study or who does not sign the informed consent
* Women of childbearing potential not using an effective method of contraception properly

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Min Bae, MD, PhD, Principal Investigator — Department of Dermatology, College of Medicine, Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Ju HJ, Kim SH, Lee JH, Kim GM, Bae JM. Efficacy and safety of tretinoin 0.05% cream to prevent hyperpigmentation during narrowband UV-B phototherapy in patients with facial vitiligo: a randomized clinical trial. J Dermatolog Treat. 2022 May;33(3):1738-1741. doi: 10.1080/09546634.2020.1817298. Epub 2020 Sep 10. PMID 32869680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a split-face trial. A single patient with paired lesions will be enrolled.
Groups:
- Left Tretinoin 0.05% Cream, Right Placebo: Tretinoin 0.05% cream (Stieva-A Cream 0.05%, 25g, GSK) on the left side of the face, moisturizer cream (Physiogel Daily Mositure Therapy Facial cream, 150mL, Stiefel) on the right side of the face for 1 month, applied once a day every night
- Left Placebo, Right Tretinoin 0.05% Cream: Tretinoin 0.05% cream (Stieva-A Cream 0.05%, 25g, GSK) on the right side of the face, moisturizer cream (Physiogel Daily Mositure Therapy Facial cream, 150mL, Stiefel) on the left side of the face for 1 month, applied once a day every night
Period: Overall Study
Arm/Group | Left Tretinoin 0.05% Cream, Right Placebo | Left Placebo, Right Tretinoin 0.05% Cream
Started | 12 | 13
Completed | 10 | 11
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Left Tretinoin 0.05% Cream, Right Placebo: The left/right sides of the face were randomly allocated to receive either topical tretinoin 0.05% (w/v) cream or moisturizer twice daily. Tretinoin 0.05% cream (Stieva-A Cream 0.05%, 25g, GSK) was applied on the half side of the face of the patients for 1 month, once a day every night.
- Left Placebo, Right Tretinoin 0.05% Cream: The left/right sides of the face were randomly allocated to receive either topical tretinoin 0.05% (w/v) cream or moisturizer twice daily. Placebo cream (Physiogel Daily Mositure Therapy Facial cream, 150mL, Stiefel) was applied on the other half side of the face of the patients for 1 month, once a day every night.
- Total: Total of all reporting groups
Arm/Group | Left Tretinoin 0.05% Cream, Right Placebo | Left Placebo, Right Tretinoin 0.05% Cream | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 13 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 12 | 13 | 25
L* value at baseline [Mean (Full Range); unit: score on a scale] — L* value (Lightness, scale from 0 to 100, based on Lab color space) measured by a spectrophotometer at baseline.
  (Higher value means lighter color.)
  score on a scale | 58.5 [51 to 64] | 56.7 [50 to 63] | 57.6 [50 to 64]

OUTCOME MEASURES:

1. Primary Outcome: The Degree of Hyperpigmentation at 12 Weeks
Description: The degree of hyperpigmentation will be assessed as L* value of Lab color space(L stands for lightness, scale from 0 to 100) using spectrophotometer at 12 weeks The higher score means the skin is lighter which means a better outcome.
Time Frame: at 12 weeks
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Left Tretinoin 0.05% Cream, Right Placebo: Tretinoin 0.05% cream (Stieva-A Cream 0.05%, 25g, GSK) applied on the left side, placebo cream on the right side of the face applied once a day every night
- Left Placebo, Right Tretinoin 0.05% Cream: Tretinoin 0.05% cream (Stieva-A Cream 0.05%, 25g, GSK) applied on the right side, placebo cream on the left side of the face applied once a day every night
Arm/Group | Left Tretinoin 0.05% Cream, Right Placebo | Left Placebo, Right Tretinoin 0.05% Cream
Number analyzed (Participants) | 10 | 11
score on a scale
  Tretinoin side | 56.8 [49 to 62] | 57.6 [52 to 63]
  Placebo side | 51.0 [46 to 60] | 54.3 [45 to 62]
Statistical Analysis 1: Comparison: Left Tretinoin 0.05% Cream, Right Placebo vs Left Placebo, Right Tretinoin 0.05% Cream; Null hypothesis: The degree of hyperpigmentation is the same between the tretinoin applied side and placebo applied side; Test type: Superiority; p = 0.002, t-test, 2 sided — P value < 0.05 was considered significant

2. Secondary Outcome: Number of Participants Who Showed ≥75% Repigmentation
Description: Number of Participants who Showed ≥75% Repigmentation assessed at 12 weeks as % change from baseline degree using VESTA as a reference value.
Time Frame: change from Baseline and at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Left Tretinoin 0.05% Cream, Right Placebo | Left Placebo, Right Tretinoin 0.05% Cream
Number analyzed (Participants) | 10 | 11
Participants
  Tretinoin side | 8 | 9
  Placebo side | 8 | 9
Statistical Analysis 1: Comparison: Left Tretinoin 0.05% Cream, Right Placebo vs Left Placebo, Right Tretinoin 0.05% Cream; Null hypothesis: The number of participants who showed ≥75% repigmentation is the same between the tretinoin applied side and placebo applied side; Test type: Superiority; p = 0.479, McNemar — P value < 0.05 was considered significant

ADVERSE EVENTS:
Time Frame: Any adverse effects (irritation, burning sensation, etc.) were collected at week 4, week 8, week 12.
Groups:
- Tretinoin 0.05% Cream Group: Tretinoin 0.05% cream 25g for 1 month, applied on the half side of the face once a day every night
  Tretinoin 0.05% cream: Stieva-A Cream 0.05%, 25g, GSK
- Placebo Cream Group: PHYSIOGEL Daily Moisture Therapy Creme 150ml for 1 month, applied on the other half of the face once a day every night
  Placebo cream: Physiogel Daily Mositure Therapy Facial cream, 150mL, Stiefel
Arm/Group | Tretinoin 0.05% Cream Group | Placebo Cream Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tretinoin 0.05% Cream Group (N=25) | Placebo Cream Group (N=25)
Irritation (Skin and subcutaneous tissue disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03933774/Prot_SAP_000.pdf